CLINICAL TRIAL: NCT01687192
Title: Multicenter Clinical Trial Evaluating the Immunological Response of Vaccination Against Infection by Human Papillomavirus (HPV) 6, 11, 16, 18 in Girls Receiving Immunosuppressive Therapy.
Brief Title: Multicenter Trial Evaluating the Immunogenicity of HPV Vaccination in Girls on Immunosuppressive Therapy.
Acronym: PRIMAVERA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CHUBX 2011/18
Record Dates: First submitted 2012-09-13; First posted 2012-09-18 (Estimated); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Transplantation; Systemic Lupus Erythematosus; Systemic Immune Disease
Keywords: Seroconversion; Immunosuppressed treatment; HPV vaccination; Immunogenicity
MeSH Terms: conditions — Lupus Erythematosus, Systemic; HIV Seropositivity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Girls and young womens receiving immunosuppressive treatment (Experimental)
  Interventions: Biological: HPV prophylactic vaccine Gardasil

INTERVENTIONS:
Biological: HPV prophylactic vaccine Gardasil — 3 injections: at Inclusion visit then 2 and 6 months after.

SUMMARY:
PRIMAVERA is a Phase IIa clinical trial, with the objective to assess the immunologic response to HPV vaccine in a population of immunocompromised girls. The principal hypothesis is that the immunologic response to tetravalent vaccine in girls who received immunosuppressive treatment is comparable to the immunologic response in girls that are not immunosuppressed.

DETAILED DESCRIPTION:
The human papillomaviruses (HPV) are the cause of the most common sexually transmitted infection. Among oncogenic HPV, HPV 16 and 18 are found in 70% of invasive cancers. Among the non-oncogenic HPV, HPV 6 and 11 are found in 90% of anogenital warts. Two prophylactic vaccines are currently available: Gardasil ® protects against HPV 6, 11, 16 and 18 and Cervarix ® that protects against HPV16 and 18. Gardasil ® is indicated for the prevention of high-grade cervical dysplasia (CIN2-3), cancers of the cervix, high-grade dysplasia of the vulva (VIN2-3) and genital warts.

The choice of Gardasil ® is linked to the theoretical risk of graft rejection with the bivalent vaccine, and the fact that the frequency of anogenital warts related to HPV 6 and 11 is increased in the immunocompromised population.

The immunosuppressed women are more likely to present abnormal cervical smears than general population.

A notice on the age of vaccination against HPV for girls to receive a transplant was made by the High Council of Public Health, recommending that vaccination against HPV could be offered to girls to benefit a transplant before the age of 14 years and according to data from the MA. The High Council of Public Health also renewed its request that studies be conducted specifically on the vaccination of girls and young women, immunocompromised, including those receiving immunosuppressive therapy.

The primary objective is to evaluate the persistence of immunological response to tetravalent HPV vaccine at 18 months after first dose of vaccine.

ELIGIBILITY:
Inclusion Criteria:

* Female gender
* Age ≥ 9 years and < 18 years
* Weight ≥ 25 kg
* Solid organ transplantation: kidney, liver, heart, lung, intestinal or combined transplant; or systemic lupus erythematosus or other systemic immune disease
* Transplantation or diagnosis of lupus or diagnosis of systemic immune disease since more than 6 months
* Immunosuppressant treatment by anti-metabolites or calcineurin inhibitors, with or without associated corticosteroids
* Minimum required period of 3 months considered as stable after transplantation or without relapse of lupus according to physician evaluation
* In case of sexual activity (assessed by auto-declaration): onset less than one year before inclusion
* Written informed consent signed by the investigator and the legal representatives of the patient, and assent by the patient

Exclusion Criteria:

* Male gender
* Pregnancy
* Age < 9 years or ≥ 18 years
* Previous HPV vaccination
* Immunosuppressive treatment by anti-TNF (adalimumab, etanercept, infliximab) or monoclonal antibodies (rituximab, anakinra, abatacept) during the last 3 months
* Active malignancy
* Active opportunistic infection
* HIV infection
* Concurrent clinical trial

Ages: 9 Years to 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 37 (Estimated)
Dates: Start 2012-10-11 (Actual); Primary Completion 2015-05 (Actual); Study Completion 2016-10-20 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate for HPV 16 and 18 at M18 | 18 months after first dose of vacinne (i.e. Inclusion visit)

SECONDARY OUTCOMES:
Geometric means of anti-HPV 6, 11, 16 and 18 antibody titers at M7, M18, and M36, respectively. | Samples collected 7, 18 and 36 months after first dose of vaccine
Proportion of patients with a good cell response at M7 and M18 | 7 and 18 months after first dose of vaccine
Proportion of patients with genital warts or cervical lesions (if relevant) | 36 months after first dose of vaccine
Number, type and time of occurrence of adverse events of any grade during 18 months after first dose of vaccine | Assessed at months 2,6,7 and 18 after first dose of vaccine

CONTACTS AND LOCATIONS:
Overall Officials: Geneviève CHENE, MD-PhD, Study Chair — University Hospital, Bordeaux, USMR; Jerome HARAMBAT, MD, Principal Investigator — University Hospital, Bordeaux
Locations (9):
- France (9):
  - CHU de Bordeaux, Hôpital Pellegrin-Enfants, Bordeaux
  - HCLyon, Hôpital Femme-mère-enfant, Bron
  - CHU de Lille, Hôpital Jeanne de Flandres, Lille
  - CHU de Montpellier, Hôpital Arnaud de Villeneuve, Montpellier
  - CHU de Nantes, Hôpital Mère-Enfants, Nantes
  - AP-HP, Hôpital Robert Debré, Paris
  - AP-HP, Hôpital Armand Trousseau, Paris
  - AP-HP, Hôpital Necker-Enfants, Paris
  - CHU de Toulouse, Hôpital des Enfants, Toulouse

REFERENCES:
- [Background] Koutsky L. The epidemiology behind the HPV vaccine discovery. Ann Epidemiol. 2009 Apr;19(4):239-44. doi: 10.1016/j.annepidem.2009.01.023. PMID 19344861
- [Background] Johnson AM, Mercer CH, Erens B, Copas AJ, McManus S, Wellings K, Fenton KA, Korovessis C, Macdowall W, Nanchahal K, Purdon S, Field J. Sexual behaviour in Britain: partnerships, practices, and HIV risk behaviours. Lancet. 2001 Dec 1;358(9296):1835-42. doi: 10.1016/S0140-6736(01)06883-0. PMID 11741621
- [Background] Winer RL, Lee SK, Hughes JP, Adam DE, Kiviat NB, Koutsky LA. Genital human papillomavirus infection: incidence and risk factors in a cohort of female university students. Am J Epidemiol. 2003 Feb 1;157(3):218-26. doi: 10.1093/aje/kwf180. PMID 12543621
- [Background] Collins S, Mazloomzadeh S, Winter H, Blomfield P, Bailey A, Young LS, Woodman CB. High incidence of cervical human papillomavirus infection in women during their first sexual relationship. BJOG. 2002 Jan;109(1):96-8. doi: 10.1111/j.1471-0528.2002.01053.x. PMID 11845815
- [Background] Myers ER, McCrory DC, Nanda K, Bastian L, Matchar DB. Mathematical model for the natural history of human papillomavirus infection and cervical carcinogenesis. Am J Epidemiol. 2000 Jun 15;151(12):1158-71. doi: 10.1093/oxfordjournals.aje.a010166. PMID 10905528
- [Background] Penn I. Occurrence of cancers in immunosuppressed organ transplant recipients. Clin Transpl. 1998:147-58. PMID 10503093
- [Background] Fairley CK, Chen S, Tabrizi SN, McNeil J, Becker G, Walker R, Atkins RC, Thomson N, Allan P, Woodburn C, et al. Prevalence of HPV DNA in cervical specimens in women with renal transplants: a comparison with dialysis-dependent patients and patients with renal impairment. Nephrol Dial Transplant. 1994;9(4):416-20. PMID 8084456
- [Background] ter Haar-van Eck SA, Rischen-Vos J, Chadha-Ajwani S, Huikeshoven FJ. The incidence of cervical intraepithelial neoplasia among women with renal transplant in relation to cyclosporine. Br J Obstet Gynaecol. 1995 Jan;102(1):58-61. doi: 10.1111/j.1471-0528.1995.tb09027.x. PMID 7833312
- [Background] Fairley CK, Sheil AG, McNeil JJ, Ugoni AM, Disney AP, Giles GG, Amiss N. The risk of ano-genital malignancies in dialysis and transplant patients. Clin Nephrol. 1994 Feb;41(2):101-5. PMID 8004825
- [Background] Kessler M, Jay N, Molle R, Guillemin F. Excess risk of cancer in renal transplant patients. Transpl Int. 2006 Nov;19(11):908-14. doi: 10.1111/j.1432-2277.2006.00383.x. PMID 17018126
- [Background] Birkeland SA, Lokkegaard H, Storm HH. Cancer risk in patients on dialysis and after renal transplantation. Lancet. 2000 May 27;355(9218):1886-7. doi: 10.1016/s0140-6736(00)02298-4. PMID 10866449
- [Background] Vajdic CM, McDonald SP, McCredie MR, van Leeuwen MT, Stewart JH, Law M, Chapman JR, Webster AC, Kaldor JM, Grulich AE. Cancer incidence before and after kidney transplantation. JAMA. 2006 Dec 20;296(23):2823-31. doi: 10.1001/jama.296.23.2823. PMID 17179459
- [Background] Nyberg G, Eriksson O, Westberg NG. Increased incidence of cervical atypia in women with systemic lupus erythematosus treated with chemotherapy. Arthritis Rheum. 1981 May;24(5):648-50. doi: 10.1002/art.1780240503. PMID 7236321
- [Background] Nath R, Mant C, Luxton J, Hughes G, Raju KS, Shepherd P, Cason J. High risk of human papillomavirus type 16 infections and of development of cervical squamous intraepithelial lesions in systemic lupus erythematosus patients. Arthritis Rheum. 2007 May 15;57(4):619-25. doi: 10.1002/art.22667. PMID 17471531
- [Background] Tam LS, Chan PK, Ho SC, Yu MM, Yim SF, Cheung TH, Wong MC, Li EK. Natural history of cervical papilloma virus infection in systemic lupus erythematosus - a prospective cohort study. J Rheumatol. 2010 Feb;37(2):330-40. doi: 10.3899/jrheum.090644. Epub 2009 Dec 23. PMID 20032093
- [Background] Kirnbauer R, Hubbert NL, Wheeler CM, Becker TM, Lowy DR, Schiller JT. A virus-like particle enzyme-linked immunosorbent assay detects serum antibodies in a majority of women infected with human papillomavirus type 16. J Natl Cancer Inst. 1994 Apr 6;86(7):494-9. doi: 10.1093/jnci/86.7.494. PMID 8133532
- [Background] Joura EA, Kjaer SK, Wheeler CM, Sigurdsson K, Iversen OE, Hernandez-Avila M, Perez G, Brown DR, Koutsky LA, Tay EH, Garcia P, Ault KA, Garland SM, Leodolter S, Olsson SE, Tang GW, Ferris DG, Paavonen J, Lehtinen M, Steben M, Bosch X, Dillner J, Kurman RJ, Majewski S, Munoz N, Myers ER, Villa LL, Taddeo FJ, Roberts C, Tadesse A, Bryan J, Lupinacci LC, Giacoletti KE, Lu S, Vuocolo S, Hesley TM, Haupt RM, Barr E. HPV antibody levels and clinical efficacy following administration of a prophylactic quadrivalent HPV vaccine. Vaccine. 2008 Dec 9;26(52):6844-51. doi: 10.1016/j.vaccine.2008.09.073. Epub 2008 Oct 16. PMID 18930097
- [Background] Garland SM, Hernandez-Avila M, Wheeler CM, Perez G, Harper DM, Leodolter S, Tang GW, Ferris DG, Steben M, Bryan J, Taddeo FJ, Railkar R, Esser MT, Sings HL, Nelson M, Boslego J, Sattler C, Barr E, Koutsky LA; Females United to Unilaterally Reduce Endo/Ectocervical Disease (FUTURE) I Investigators. Quadrivalent vaccine against human papillomavirus to prevent anogenital diseases. N Engl J Med. 2007 May 10;356(19):1928-43. doi: 10.1056/NEJMoa061760. PMID 17494926
- [Background] FUTURE II Study Group. Quadrivalent vaccine against human papillomavirus to prevent high-grade cervical lesions. N Engl J Med. 2007 May 10;356(19):1915-27. doi: 10.1056/NEJMoa061741. PMID 17494925
- [Background] Mao C, Koutsky LA, Ault KA, Wheeler CM, Brown DR, Wiley DJ, Alvarez FB, Bautista OM, Jansen KU, Barr E. Efficacy of human papillomavirus-16 vaccine to prevent cervical intraepithelial neoplasia: a randomized controlled trial. Obstet Gynecol. 2006 Jan;107(1):18-27. doi: 10.1097/01.AOG.0000192397.41191.fb. PMID 16394035
- [Background] Villa LL, Costa RL, Petta CA, Andrade RP, Ault KA, Giuliano AR, Wheeler CM, Koutsky LA, Malm C, Lehtinen M, Skjeldestad FE, Olsson SE, Steinwall M, Brown DR, Kurman RJ, Ronnett BM, Stoler MH, Ferenczy A, Harper DM, Tamms GM, Yu J, Lupinacci L, Railkar R, Taddeo FJ, Jansen KU, Esser MT, Sings HL, Saah AJ, Barr E. Prophylactic quadrivalent human papillomavirus (types 6, 11, 16, and 18) L1 virus-like particle vaccine in young women: a randomised double-blind placebo-controlled multicentre phase II efficacy trial. Lancet Oncol. 2005 May;6(5):271-8. doi: 10.1016/S1470-2045(05)70101-7. PMID 15863374
- [Background] Ault KA; Future II Study Group. Effect of prophylactic human papillomavirus L1 virus-like-particle vaccine on risk of cervical intraepithelial neoplasia grade 2, grade 3, and adenocarcinoma in situ: a combined analysis of four randomised clinical trials. Lancet. 2007 Jun 2;369(9576):1861-1868. doi: 10.1016/S0140-6736(07)60852-6. PMID 17544766
- [Background] Joura EA, Leodolter S, Hernandez-Avila M, Wheeler CM, Perez G, Koutsky LA, Garland SM, Harper DM, Tang GW, Ferris DG, Steben M, Jones RW, Bryan J, Taddeo FJ, Bautista OM, Esser MT, Sings HL, Nelson M, Boslego JW, Sattler C, Barr E, Paavonen J. Efficacy of a quadrivalent prophylactic human papillomavirus (types 6, 11, 16, and 18) L1 virus-like-particle vaccine against high-grade vulval and vaginal lesions: a combined analysis of three randomised clinical trials. Lancet. 2007 May 19;369(9574):1693-702. doi: 10.1016/S0140-6736(07)60777-6. PMID 17512854
- [Background] Hildesheim A, Herrero R, Wacholder S, Rodriguez AC, Solomon D, Bratti MC, Schiller JT, Gonzalez P, Dubin G, Porras C, Jimenez SE, Lowy DR; Costa Rican HPV Vaccine Trial Group. Effect of human papillomavirus 16/18 L1 viruslike particle vaccine among young women with preexisting infection: a randomized trial. JAMA. 2007 Aug 15;298(7):743-53. doi: 10.1001/jama.298.7.743. PMID 17699008
- [Background] Slade BA, Leidel L, Vellozzi C, Woo EJ, Hua W, Sutherland A, Izurieta HS, Ball R, Miller N, Braun MM, Markowitz LE, Iskander J. Postlicensure safety surveillance for quadrivalent human papillomavirus recombinant vaccine. JAMA. 2009 Aug 19;302(7):750-7. doi: 10.1001/jama.2009.1201. PMID 19690307
- [Background] Villa LL, Costa RL, Petta CA, Andrade RP, Paavonen J, Iversen OE, Olsson SE, Hoye J, Steinwall M, Riis-Johannessen G, Andersson-Ellstrom A, Elfgren K, Krogh Gv, Lehtinen M, Malm C, Tamms GM, Giacoletti K, Lupinacci L, Railkar R, Taddeo FJ, Bryan J, Esser MT, Sings HL, Saah AJ, Barr E. High sustained efficacy of a prophylactic quadrivalent human papillomavirus types 6/11/16/18 L1 virus-like particle vaccine through 5 years of follow-up. Br J Cancer. 2006 Dec 4;95(11):1459-66. doi: 10.1038/sj.bjc.6603469. Epub 2006 Nov 21. PMID 17117182
- [Background] Olsson SE, Villa LL, Costa RL, Petta CA, Andrade RP, Malm C, Iversen OE, Hoye J, Steinwall M, Riis-Johannessen G, Andersson-Ellstrom A, Elfgren K, von Krogh G, Lehtinen M, Paavonen J, Tamms GM, Giacoletti K, Lupinacci L, Esser MT, Vuocolo SC, Saah AJ, Barr E. Induction of immune memory following administration of a prophylactic quadrivalent human papillomavirus (HPV) types 6/11/16/18 L1 virus-like particle (VLP) vaccine. Vaccine. 2007 Jun 21;25(26):4931-9. doi: 10.1016/j.vaccine.2007.03.049. Epub 2007 Apr 20. PMID 17499406
- [Background] Reisinger KS, Block SL, Lazcano-Ponce E, Samakoses R, Esser MT, Erick J, Puchalski D, Giacoletti KE, Sings HL, Lukac S, Alvarez FB, Barr E. Safety and persistent immunogenicity of a quadrivalent human papillomavirus types 6, 11, 16, 18 L1 virus-like particle vaccine in preadolescents and adolescents: a randomized controlled trial. Pediatr Infect Dis J. 2007 Mar;26(3):201-9. doi: 10.1097/01.inf.0000253970.29190.5a. PMID 17484215
- [Background] Levin MJ, Moscicki AB, Song LY, Fenton T, Meyer WA 3rd, Read JS, Handelsman EL, Nowak B, Sattler CA, Saah A, Radley DR, Esser MT, Weinberg A; IMPAACT P1047 Protocol Team. Safety and immunogenicity of a quadrivalent human papillomavirus (types 6, 11, 16, and 18) vaccine in HIV-infected children 7 to 12 years old. J Acquir Immune Defic Syndr. 2010 Oct;55(2):197-204. doi: 10.1097/QAI.0b013e3181de8d26. PMID 20574412
- [Background] Grabowska K, Wang X, Jacobsson A, Dillner J. Evaluation of cost-precision rations of different strategies for ELISA measurement of serum antibody levels. J Immunol Methods. 2002 Dec 20;271(1-2):1-15. doi: 10.1016/s0022-1759(02)00334-4. PMID 12445724
- [Background] Dessy FJ, Giannini SL, Bougelet CA, Kemp TJ, David MP, Poncelet SM, Pinto LA, Wettendorff MA. Correlation between direct ELISA, single epitope-based inhibition ELISA and pseudovirion-based neutralization assay for measuring anti-HPV-16 and anti-HPV-18 antibody response after vaccination with the AS04-adjuvanted HPV-16/18 cervical cancer vaccine. Hum Vaccin. 2008 Nov-Dec;4(6):425-34. doi: 10.4161/hv.4.6.6912. Epub 2008 Nov 11. PMID 18948732
- [Background] Waterboer T, Sehr P, Michael KM, Franceschi S, Nieland JD, Joos TO, Templin MF, Pawlita M. Multiplex human papillomavirus serology based on in situ-purified glutathione s-transferase fusion proteins. Clin Chem. 2005 Oct;51(10):1845-53. doi: 10.1373/clinchem.2005.052381. Epub 2005 Aug 11. PMID 16099939
- [Background] Michael KM, Waterboer T, Sehr P, Rother A, Reidel U, Boeing H, Bravo IG, Schlehofer J, Gartner BC, Pawlita M. Seroprevalence of 34 human papillomavirus types in the German general population. PLoS Pathog. 2008 Jun 20;4(6):e1000091. doi: 10.1371/journal.ppat.1000091. PMID 18566657
- [Background] Mendez F, Munoz N, Posso H, Molano M, Moreno V, van den Brule AJ, Ronderos M, Meijer C, Munoz A; Instituto Nacional de Cancerologia Human Papillomavirus Study Group. Cervical coinfection with human papillomavirus (HPV) types and possible implications for the prevention of cervical cancer by HPV vaccines. J Infect Dis. 2005 Oct 1;192(7):1158-65. doi: 10.1086/444391. Epub 2005 Aug 29. PMID 16136457